CLINICAL TRIAL: NCT04391049
Title: Phase I Trial With Expansion Cohort of OBP-301 (Telomelysin™) and Definitive Chemoradiation for Patients With Locally Advanced Esophageal and Gastroesophageal Cancer Who Are Not Candidates for Surgery
Brief Title: Testing the Addition of the Anti-cancer Viral Therapy Telomelysin™ to Chemoradiation for Patients With Advanced Esophageal Cancer and Are Not Candidates for Surgery
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GI007; NCI-2020-02320 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GI007 (Other: NRG Oncology); NRG-GI007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Esophageal Adenocarcinoma; Advanced Gastroesophageal Junction Adenocarcinoma; Clinical Stage II Esophageal Adenocarcinoma AJCC v8; Clinical Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IIA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IIB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage II Esophageal Adenocarcinoma AJCC v8; Pathologic Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage II Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage II Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Unresectable Gastroesophageal Junction Adenocarcinoma; Squamous Cell Carcinoma; Squamous Cell Cancer
Keywords: OBP-301; viral therapy
MeSH Terms: conditions — Carcinoma, Squamous Cell; Neoplasms, Squamous Cell | interventions — Carboplatin; Paclitaxel; Taxes; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (OBP-301, carboplatin, paclitaxel, radiation) (Experimental): Patients receive OBP-301 (1×10^12 vp/mL) by intra-tumoral injection via endoscopy on days -3, 12, and 26. Patients also receive paclitaxel IV (50 mg/m^2) over 60 minutes followed by carboplatin IV (AUC 2) over 30 minutes and on days 1, 8, 15, 22, and 29, and undergo radiation therapy (1.8 Gy/faction) on Monday through Friday beginning day 1 for 28 fractions (50.4 Gy total) over 5.5 weeks. All treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiation Therapy; Biological: Telomerase-specific Type 5 Adenovirus OBP-301

INTERVENTIONS:
Drug: Carboplatin — Intravenously (IV)
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Paclitaxel — Intravenously (IV)
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Radiation: Radiation Therapy — Daily fractions
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
Biological: Telomerase-specific Type 5 Adenovirus OBP-301 — Intra-tumoral injection
  Other Names: OBP-301; Telomelysin ™

SUMMARY:
This phase I trial studies the side effects of OBP-301 when given together with carboplatin, paclitaxel, and radiation therapy in treating patients with esophageal or gastroesophageal cancer that invades local or regional structures. OBP-301 is a virus that has been designed to infect and destroy tumor cells (although there is a small risk that it can also infect normal cells). Chemotherapy drugs, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving OBP-301 with chemotherapy and radiation therapy may work better than standard chemotherapy and radiation therapy in treating patients with esophageal or gastroesophageal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the addition of OBP-301 to chemoradiation with carboplatin/paclitaxel is safe.

SECONDARY OBJECTIVES:

I. To assess toxicities associated with the addition of OBP-301 to chemoradiation.

II. To assess the number of clinical complete responses (cCR).

III. To assess the number of patients alive/without progression (progression-free survival [PFS]) and the number of patients alive (overall survival [OS]) at 1 and 2 years.

EXPLORATORY OBJECTIVE:

I. To report correlate outcomes - cCR, PFS and OS - with immune and virus-based correlative assays.

OUTLINE:

This study will evaluate an initial dose of OBP-301 and a de-escalated dose, if needed.

Patients receive OBP-301 by intratumoral injection via endoscopy on days -3, 12, and 26. Patients also receive carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 60 minutes on days 1, 8, 15, 22, and 29, and undergo radiation therapy on Monday through Friday beginning day 1 for 28 fractions over 5.5 weeks. All treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 6-8 weeks, then every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of adenocarcinoma or squamous cell carcinoma (SCC) of the esophagus or gastroesophageal junction (GEJ) within 90 days prior to registration

  * Gastroesophageal junction tumors must be Siewert type I/II
* Required diagnostic workup for study entry:

  * History/physical examination prior to registration
  * Computed tomography (CT) of the chest/abdomen with intravenous contrast within 28 days prior to registration; If CT contrast is contraindicated magnetic resonance imaging (MRI) of the chest/abdomen without contrast is permitted
  * Bronchoscopy for squamous cell carcinoma (SCC) tumors that are adjacent to the airway to exclude a tracheoesophageal fistula within 42 days prior to registration
  * Endoscopic ultrasound (if technically feasible) within 90 days prior to registration
  * Whole body positron emission tomography (PET)/CT scan within 42 days prior to registration: Note: scan will be used for radiation treatment planning, in addition to ruling out metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 within 14 days prior to registration
* Adequate hematologic function within 14 days prior to registration defined as follows Absolute neutrophil count ≥ 1,500/mcL (within 14 days prior to registration) Hemoglobin ≥ 9 gm/dL (within 14 days prior to registration) Platelets ≥ 100,000/mcL (within 14 days prior to registration)
* Adequate renal function within 14 days prior to registration defined as follows Creatinine clearance of ≥ 50 ml/min (as calculated by Cockcroft-Gault equation) (within 14 days prior to registration)
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (within 14 days prior to registration)
* AST/ALT ≤ 2.5 x ULN
* Patients for whom non-operative management is a viable option in the opinion of a thoracic surgeon and/or multidisciplinary team and are candidates for chemoradiation; this does not preclude patients from receiving surgery after chemoradiation if felt to me medically indicated;
* Patients must, in the opinion of a treating gastroenterologist, have a tumor that is amenable to intratumoral injection with at least 1 mL (1 x 10^12 vp/mL) of OBP-301 and be a candidate for 3 endoscopy procedures
* Female patients of child bearing potential must have a negative serum/urine pregnancy test within 14 days prior to study entry. A female not of childbearing potential is one who has undergone a hysterectomy, bilateral oophorectomy, tubal ligation, or who has had no menses for 12 consecutive months
* Patients of reproductive potential must agree to use effective contraception for the duration of study treatment as well as 6 months (for women) or 12 months (for men) after the last administered injection of OBP-301. Effective contraception includes oral contraceptives, implantable hormonal contraception, double-barrier method or intrauterine device
* The patient must provide study-specific informed consent prior to study entry
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Known acute or chronic hepatitis B or C infection (testing not required prior to study entry in patients with no known history of hepatitis B or C)

  * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
  * For patients with a history of hepatitis C virus (HCV) infection, they must (i) have been treated and cured, (ii) for patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months prior to study entry are eligible for this trial

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease including:

  * Positive malignant cytology of the pleura, pericardium or peritoneum
  * Radiographic evidence of involvement of any adjacent mediastinal structure, e.g. aorta, trachea, which would increase the risk of repeated endoscopic interventions
  * Tracheoesophageal fistula
  * Radiographic evidence of distant organ involvement
  * Non-regional lymph nodes that cannot be contained within a radiation field
* More than 1 esophageal lesion
* Prior systemic chemotherapy for the study cancer
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Biopsy-proven tumor invasion of the tracheobronchial tree or presence of tracheoesophageal fistula or recurrent laryngeal or phrenic nerve paralysis
* For patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, a New York Heart Association functional classification 2C or worse
* Uncontrolled diabetes
* Infection requiring IV antibiotics at the time of registration
* Patients requiring immunosuppressive medications including chronic suppressive steroid therapy (greater than the equivalent of 20 mg/day of prednisone), methotrexate, azathioprine and TNF-alpha blockers within 7 days prior to study entry
* Received live vaccine within 30 days prior to registration
* Received a blood transfusion, hematopoietic agent; granulocyte-colony stimulating factor (G-CSF), and/or oxygen supplementation within 7 days before the screening lab
* Breast feeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2026-10-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Y Ku, Principal Investigator — NRG Oncology
Locations (17):
- United States (17):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants who started treatment.
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 74 [62 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Zubrod Performance Status [Count of Participants; unit: Participants]
  0 (Asymptomatic) | 6
  1 (Symptomatic but completely ambulatory) | 9
Histologic Type [Count of Participants; unit: Participants] — A description of a tumor based on how the cancer cells and tissue look under a microscope.
  Participants
    Adenocarcinoma | 11
    Squamous cell carcinoma | 4
Tumor Location [Count of Participants; unit: Participants]
  Esophagogastric junction | 3
  Esophagus | 12
Siewert Type for Esophagogastric Junction [Count of Participants; unit: Participants] — "Siewert type" refers to a classification system used to categorize tumors located at the gastroesophageal junction (GEJ) based on the location of the tumor's epicenter relative to the GEJ, with Type I being tumors located 1-5cm above the GEJ, Type II at the GEJ itself (within 1cm above and 2cm below), and Type III being tumors located 2-5cm below the GEJ; essentially indicating whether the tumor originated more from the esophagus (Type I) or stomach (Type III) with Type II being considered the true GEJ cancer. Population: Participants with tumor location of esophagogastric junction.
  Participants
    number analyzed (Participants) | 3
    Type I | 2
    Type II | 1
Clinical T Category [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 8th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail.
  Participants
    T1b (Tumor has invaded the submucosa, but not penetrated the muscularis propria.) | 2
    T2 (Tumor invades the muscularis propria.) | 4
    T3 (Tumor invades the adventitia.) | 9
Clinical N Category [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 8th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. A higher number means the cancer is in more lymph nodes, farther away from the original tumor.
  Participants
    N0 (No regional lymph nodes) | 3
    N1 (1-2 regional lymph nodes) | 7
    N2 (3-6 regional lymph nodes) | 2
    N3 (7 or more regional lymph nodes) | 2
    NX (Regional lymph nodes cannot be assessed or evaluated) | 1
Extent of Dysphagia [Count of Participants; unit: Participants] — Dysphagia, or difficulty swallowing, can range from mild to severe, and can affect a person's ability to eat and drink. The extent of dysphagia can depend on the underlying cause and the severity of the condition.
  Participants
    Asymptomatic | 5
    Symptomatic, unrestricted diet | 5
    Symptomatic, soft foods only | 4
    Symptomatic, liquids only | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Any Dose-Limiting Toxicities (DLTs)
Description: Adverse events are graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, which grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. A DLT is defined as the following that are definitely or probably attributed to OBP-301:
  * Any grade ≥3 adverse event EXCEPT for the following:
    * Grade 3 nausea/vomiting
    * Grade 3 esophagitis or dehydration
    * The first occurrence of grade 3/4 neutropenia
    * Grade 3/4 lymphopenia (since this is a known toxicity of chemoradiation and OBP-301)
  * Any toxicity that leads to a >14-day cumulative delay in chemoradiation.
  If 0 or 1 participants of 6 participants experienced a DLT, then the treatment regimen would be considered safe (and 9 more would be accrued for secondary endpoints). Otherwise, the regimen would be deemed too toxic and a second cohort of six participants would be accrued to a lower dose of OBP-301 (1 x 10^11 vp/mL).
Time Frame: From start of protocol treatment until 30 days after the completion of chemoradiation, approximately 10 weeks.
Population: First six eligible participants who started all protocol treatment and either experienced a DLT in the evaluation period or completed the evaluation period without a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
Number analyzed (Participants) | 6
Participants | 0

2. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: The Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From start of protocol treatment to last follow-up. Maximum follow-up was 28.7 months.
Population: Eligible participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
Number analyzed (Participants) | 15
Participants
  All adverse events: None reported | 0
  All adverse events: Grade 1 | 1
  All adverse events: Grade 2 | 1
  All adverse events: Grade 3 | 7
  All adverse events: Grade 4 | 4
  All adverse events: Grade 5 | 2
  Definitely or probably related to any protocol treatment: None reported | 1
  Definitely or probably related to any protocol treatment: Grade 1 | 3
  Definitely or probably related to any protocol treatment: Grade 2 | 1
  Definitely or probably related to any protocol treatment: Grade 3 | 8
  Definitely or probably related to any protocol treatment: Grade 4 | 1
  Definitely or probably related to any protocol treatment: Grade 5 | 1
  Definitely or probably related to OBP-301 protocol treatment: None reported | 7
  Definitely or probably related to OBP-301 protocol treatment: Grade 1 | 2
  Definitely or probably related to OBP-301 protocol treatment: Grade 2 | 5
  Definitely or probably related to OBP-301 protocol treatment: Grade 3 | 0
  Definitely or probably related to OBP-301 protocol treatment: Grade 4 | 1
  Definitely or probably related to OBP-301 protocol treatment: Grade 5 | 0

3. Secondary Outcome: Number of Participants With Clinical Complete Response (cCR)
Description: Clinical complete response is defined as grossly free of disease as determined by a visual inspection or if the visual inspection was not certain, then a negative biopsy. The number of participants is determined for two populations:
  * Complete case analysis only includes eligible participants who started protocol treatment and were assessed for cCR;
  * Sensitivity analysis includes all eligible participants who started protocol treatment and counts participants without an assessment as not achieving a cCR.
Time Frame: 6-8 weeks after completion of chemoradiation, approximately 11.5-13.5 weeks from baseline.
Population: Eligible and started protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
Number analyzed (Participants) | 15
Participants
  Complete Case Analysis: number analyzed (Participants) | 13
  Complete Case Analysis | 13
  Sensitivity Analysis | 13

4. Secondary Outcome: Number of Participants Alive Without Progression at 1 and 2 Years
Description: Progression is defined as pathologically confirmed recurrence of local disease or clinical evidence of distant disease.
Time Frame: At 1 and 2 years
Reporting Status: Not Posted, anticipated posting 2026-10

5. Secondary Outcome: Number of Participants Alive at 1 and 2 Years
Time Frame: At 1 and 2 years
Reporting Status: Not Posted, anticipated posting 2026-10

ADVERSE EVENTS:
Time Frame: From start of protocol treatment to last follow-up. Maximum follow-up was 28.7 months.
Description: All-cause mortality and adverse events were assessed in eligible participants who started protocol treatment.
Arm/Group | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation)
All-Cause Mortality (participants affected / at risk) | 5/15
Serious Adverse Events (participants affected / at risk) | 7/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation) (N=15)
Atrial fibrillation (Cardiac disorders) | 1
Esophageal fistula (Gastrointestinal disorders) | 1
Esophageal stenosis (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (OBP-301, Carboplatin, Paclitaxel, Radiation) (N=15)
Anemia (Blood and lymphatic system disorders) | 10
Eosinophilia (Blood and lymphatic system disorders) | 2
Sinus tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Belching (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 3
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 5
Esophageal ulcer (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 5
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 13
Fever (General disorders) | 4
Flu like symptoms (General disorders) | 2
Gait disturbance (General disorders) | 1
General disorders and administration site conditions - Other (General disorders) | 1
Injection site reaction (General disorders) | 1
Localized edema (General disorders) | 1
Malaise (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Esophageal infection (Infections and infestations) | 1
Infections and infestations - Other (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Creatinine increased (Investigations) | 2
Investigations - Other (Investigations) | 1
Lymphocyte count decreased (Investigations) | 12
Neutrophil count decreased (Investigations) | 9
Platelet count decreased (Investigations) | 8
Thyroid stimulating hormone increased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 1
Glucosuria (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Flushing (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 4
Thromboembolic event (Vascular disorders) | 2
Vascular disorders - Other (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04391049/Prot_SAP_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT04391049/ICF_001.pdf